CLINICAL TRIAL: NCT03293186
Title: Anti-adhesive Effect and Safety of "Thermo-sensitive Adhesion Barrier (MEDICLORE)" by Using Double-blind Test in Thyroid Surgery
Brief Title: Anti-adhesive Effect and Safety of "Thermo-sensitive Adhesion Barrier (MEDICLORE)"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su-jin Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SNUHthyroid2
Record Dates: First submitted 2017-08-18; First posted 2017-09-26 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Adhesion; Thyroidectomy
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use MEDICLORE (Experimental): use mediclore at the end of surgery
  Interventions: Combination Product: MEDICLORE
- No antiadhesive product (No Intervention): use no antiadhesive product at the end of surgery

INTERVENTIONS:
Combination Product: MEDICLORE — use MEDICLORE at the end of surgery as antiadhesive product
  Arms: Use MEDICLORE

SUMMARY:
One of most important complication of thyroid surgery is adhesion. There are many anti-adhesive materials, but none of them showed significant outcomes. The investigators planned double blind prospective study of "Thermo-sensitive Adhesion Barrier (MEDICLORE)" to reveal anti-adhesive effect of MEDICLORE. The investigators will recruit total 90 patients (control group 45, experimental group 45) and compare postoperative outcomes about adhesion.

ELIGIBILITY:
Inclusion Criteria:

* planned to perform thyroidectomy due to thyroid nodule
* no evidence of distant metastasis or invasion to adjacent organ in thyroid cancer
* normal preoperative vocal cord movement
* normal preoperative laboratory study

Exclusion Criteria:

* uncontrolled hypertension, diabetes, chronic renal failure, coagulopathy
* history of keloid or hypertrophic scar
* Graves disease or hashimoto thyroiditis patients
* aspirin or anticoagulant medication within 7 days
* radiation exposure to the head and neck
* previous operation to the neck
* history of allergic reaction to drugs
* pregnant women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of postoperative adhesion will checked using answer of questionnaire that participants and physicians replied. | Participants will be followed from the operation to postoperative 2weeks, 3months, 6months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No